CLINICAL TRIAL: NCT03427307
Title: Association of Lipopolysaccharide-binding Protein (LBP) and Atherosclerotic Vascular Disease in Taiwanese Hemodialysis Patients
Brief Title: Serum Level of Lipopolysaccharide-binding Protein (LBP) and Atherosclerosis in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 106064
Record Dates: First submitted 2018-01-27; First posted 2018-02-09 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: Lipopolysaccharide-binding protein; inflammation; ASCVD
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background In hemodialysis (HD) patients, impaired gut barrier and alteration in microbiota in the gut is thought to increase the risk of bacterial translocation and chronic inflammation. Lipopolysaccharide-binding protein (LBP) is an acute-phase reactant that mediates immune responses triggered by microbial products. Our aim is to investigate the relationship between circulating levels of LBP, inflammatory markers and incident atherosclerotic vascular events in HD patients and follow-up this defined cohort for 3 years.

Methods A total of 300 HD patients will be recruited. The LBP and inflammatory markers will be determined using immuoassay methods annually. A bioimpedance spectroscopy device will used for body fat composition measurement and measurements will be done annually. Arterial stiffness is evaluated by measuring PWV in the heart-femoral segment using an automatic waveform analyzer.

DETAILED DESCRIPTION:
Study Design and Population

Patient Population

To be included in the study, patients have to be at least 20-years-old and on outpatient hemodialysis (HD) for at least 3 months. Patients are excluded if they had an acute infection or malignancy. A total of 360 long-term HD patients are randomly invited and agreed to participate in the study. The medical record is thoroughly reviewed for each subject by a collaborating physician in the study. Information such as underlying kidney disease, cardiovascular disease history, and other comorbid illnesses will be abstracted.

Study Parameters

Predialysis blood samples are obtained on a mid-week day. Within 30 min after sampling, the remaining blood is centrifuged at 3,000 g for 10 min, immediately aliquoted and frozen at -70°C until further analysis. Total serum cholesterol is measured through the reaction of cholesterol esterase/cholesterol oxidase/peroxidase, using Hitachi 747 (Hitachi, Bohemia, NY, USA). HDL cholesterol is quantified after precipitation with polyethylene glycol at room temperature. Serum glucose concentrations are measured by the glucose oxidase method. Low-density lipoprotein cholesterol is calculated using the Friedewald formula. Total serum triglycerides are measured through the reaction of glycerol/phosphate/oxidase and peroxidase. The serum levels of high-sensitivity C-reactive protein (hsCRP) are measured using a Behring Nephelometer II (Dade Behring, Tokyo, Japan). Plasma levels of Interleukin-6 (IL-6) and soluble CD14(sCD14) are measured by a commercially available enzyme linked immunosorbent assay (ELISA) (Quantikine HS Immunoassay kit, R&D System, Minneapolis, MN). Concentrations Interleukin-6(IL-10), and Tumor necrosis factor-alpha(TNF-α) are simultaneously determined by the Multiplex® (R&D Systems, Minnesota, MN, USA). Serum levels of LBP will be measured using a commercial enzyme-linked immunosorbent assay (HK315-02, HyCult Biotech Inc., Uden, the Netherlands) as per manufacturer's instructions. The intra- and inter-assay coefficients of LBP variation are <5 and <10%, respectively. Besides, serum from 40 normal control subjects will be used for interassay variation. Both the intra- and the interassay coefficients of variation were <8.0%. All samples will be measured in duplicates and the mean value is reported in μg/mL

Percent fat is measured with Bioelectric Impedance Spectroscopy

Whole-body bioelectric impedance spectroscopy (BIS) measurement using a body composition monitor (BCM: Fresenius Medical Care, Bad Homburg, Germany) is performed on each of the participants enrolled in the study as described previously [28]. Briefly, measurements were taken on the day before dialysis with the patient calm, supine, and relaxed in the dialysis bed for 10 minutes. Four electrodes were placed on the patient's hand and foot on the side contra lateral to their arteriovenous fistula. The basic principle of this machine is the use of the bioimpedance spectroscopy which determines the fluid content of the body by measuring the serial values of electric impedance by applying small microAmp electric currents at 50 different frequencies between 5 and 1000 kHz. These impedance data are used to obtain the amount of total body water, intracellular water and extracellular water through a special fluid model and information about other body compositions, such as fat tissue or lean tissue, through a physiological body composition model [29]. The major estimates the body composition measured by BCM-BIS are as follows: (1) lean tissue mass (LTM -mainly muscle), fat mass (FAT), and adipose tissue mass (ATM-mainly fat with its relevant hydration)

Measurement of arterial stiffness

Arterial stiffness is evaluated by measuring PWV in the heart-femoral segment using an automatic waveform analyzer.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes aged between 20-90 years.
2. Received stable hemodialysis at least 3 months.
3. Written informed consent.

Exclusion Criteria:

1. patients with severe infections, severe heart disease and liver disease, malignancy, autoimmune disorders, severe malnutrition, or clinical conditions requiring oral nutrition supplements;
2. Inability to follow protocol.
3. Pregnancy or wishing/trying to get pregnant

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients have to be at least 20-years-old and on outpatient hemodialysis (HD) for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2018-06-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Atherosclerotic events | 3 years
  Incident atherosclerotic vascular events in HD patients

SECONDARY OUTCOMES:
All-cause mortality | 3 years
  The association of LBP with all-cause mortality
Association with inflammatory markers | 3 years
  TNF-alpha, Interleukin-10(IL-10), Interleukin-6 (IL-6) and soluble (sCD14) are measured using an enzyme-linked immunosorbent assay (ELISA) annually

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan